CLINICAL TRIAL: NCT06749964
Title: Cancer-related Pain and Associated Difficulties: Using Ecological Momentary Assessment and N-of-1 Trial Methods to Adapt and Pilot Test an Internet-delivered CBT Program Based on the Psychological Flexibility Model of Chronic Pain
Brief Title: An N-of-1 Trial of an Internet-delivered CBT Program Based on the Psychological Flexibility Model of Chronic Pain for Cancer-related Difficulties
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Swedish Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-04724-01
Record Dates: First submitted 2024-12-11; First posted 2024-12-27 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Chronic Cancer-related Pain
Keywords: chronic cancer-related pain; psychological flexibility; internet delivered cognitive behavioral therapy; n-of-1 design; mediation
MeSH Terms: conditions — Negotiating

STUDY DESIGN:
Intervention Model Description: This study applies a nonconcurrent, randomised baseline length, single case experimental design (SCED) where each participant serves as their own control. Participants are randomized to a 7 - 21 days long Baseline Phase wherein they receive no intervention, immediately followed by the 5-week Treatment Phase, and then a 3-month Follow-Up Phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain focused CBT for chronic pain (Experimental): Baseline consists of a random assigned period between 7 and 21 days with measurements and no intervention.
  Intervention consists of 8 sessions of psychological flexibility training over 5 weeks.
  Interventions: Behavioral: Internet-delivered, therapist-assisted, pain-focused CBT based on the psychological flexibility model for chronic pain

INTERVENTIONS:
Behavioral: Internet-delivered, therapist-assisted, pain-focused CBT based on the psychological flexibility model for chronic pain — 8-session intervention, twice weekly for the first 3 weeks and once weekly for the final 2 weeks (45-60 min each session) aimed at promoting psychological flexibility. Treatment involves a mixture of video and audiotaped presentations and homework activities for the participant.

SUMMARY:
Chronic pain is a commonly occurring complication of cancer and can have negatively impact day-to-day functioning and well-being. The recommended treatment for all forms of chronic pain is cognitive behavioral therapy (CBT). However, access to this treatment in primary and specialist care is limited, including access to specialist pain clinics that do not routinely accept people with cancer-related pain. In addition, we know from clinical trials of pain-focused CBT that the symptom presentation of patients can vary greatly and may require interventions that are more tailored to their specific needs.

The primary objective of the research is to test the feasibility, acceptability and preliminary efficacy of an internet-delivered, therapist-assisted, intervention for chronic pain with adults suffering from chronic cancer-related pain. The intervention is a form of CBT called Acceptance Commitment Therapy (ACT) and is based on the psychological flexibility model of pain. Psychological flexibility refers to an overall pattern of persistent behaviors characterized by a present-moment focus, acceptance rather than avoidance of distressing symptoms, and engagement with one's core values and goals. The intervention aims to improve overall functioning and well-being by helping participants to develop persistent patterns of behavior that align with with their core values and goals (e.g., personal, family, social, health, occupational) despite the presence of pain and other distressing symptoms.

To achieve this aim, an existing pain-focused, internet-delivered, psychological flexibility based intervention was modified specifically for cancer-related pain with input from cancer patients and survivors. The 8-session, online intervention involves a mixture of written, audio, and videotaped materials, and instructions for experiential exercises, all of which are designed to reduce unhelpful coping behaviors and to increase psychological flexibility. Participants receive written support (and ask questions) from a therapist via the online platform where the intervention is hosted. Where necessary, participants may also access a limited number of face-to-face meetings (online) with their therapist. During the treatment phase, information from daily diary recordings (via smartphone) are used to provide individualized support to participants in the form of text messages from a therapist via the online platform. Where necessary, a limited number of face-to-face sessions (online) with a therapist are scheduled.

DETAILED DESCRIPTION:
The number of long-term cancer survivors is steadily increasing due to advances in early detection and treatment. At the same time, the number of cancer patients and survivors requiring treatment for complications of cancer is also increasing. Among the most common of these complications is chronic pain, defined as pain that persists for three or more months, and that develops either as a consequence of the disease or its treatments. Chronic cancer-related pain is associated with an increased risk of fatigue, emotional distress, occupational difficulties, increased healthcare usage, and needing assistance with activities of daily living. There are now a variety of medications that can be prescribed during cancer treatment or palliative care to reduce acute pain. However, longer-term use of these medications for chronic pain brings an increased risk of other health and behavioral difficulties. International guidelines recommend cognitive behavioural therapy (CBT) for chronic pain. However, it is widely recognized that chronic pain in cancer patients and survivors is under treated in primary and specialist care settings. This is partly due to the limited availability of therapists who can provide pain-focused CBT programs and specialist pain rehabilitation clinics not routinely accepting individuals with cancer-related pain.

One evidence-based and recommended variant of CBT for chronic pain is Acceptance and Commitment Therapy (ACT). ACT works to increase "psychological flexibility" through experiential exercises focused on developing a present-moment focus (mindfulness), openness to rather than avoidance of distressing symptoms, awareness of one's core values and goals, and commitment to behaving in line with these values/goals. Studies have found that cancer patients and survivors who are higher in psychological flexibility have greater overall well-being and functioning despite the presence of chronic cancer-related pain and associated difficulties. However, there is as yet limited research investigating the efficacy of ACT for cancer-related pain.

Given the large and increasing number of individuals diagnosed with cancer each year, and that up to 40% will develop chronic cancer-related pain, there is a need for effective treatments that can be accessed outside of specialist pain clinics. Digitally delivered interventions, either via smartphones, computers or teleconferencing, often collectively referred to as mobile-health interventions (mHealth), are seen as a cost-effective method for increasing access treatments for individuals with pain arising from diverse difficulties, including cancer. Also, there is now widespread recognition that to improve the efficacy of pain-focused CBT, clinicians and researchers need to develop methods for personalizing the treatment interventions to better reflect the variety of clinical presentations of pain patients.

The main objective of this study is to test the feasibility, acceptability, and preliminary efficacy of an internet-delivered, therapist-assisted, ACT intervention for adults suffering from chronic cancer-related pain and associated difficulties. Specifically, the investigators aim to test:

1. whether the intervention is feasible and acceptable;
2. using each participant as their own control, to test the efficacy of the intervention for the primary (pain interference) and secondary outcomes (pain intensity, fatigue, fear of cancer recurrence, depression, anxiety, overall functioning, well-being, and psychological flexibility) at the individual and group level;
3. whether treatment gains are maintained at a 3-month follow-up; and
4. whether outcomes are mediated by changes in psychological flexibility.

To achieve the project's goals, a non-concurrent, randomized, multiple-baseline across participants, single case experimental design will be used. During the baseline and treatment phases, participants complete twice-daily recording of symptoms, functioning and psychological flexibility via a smartphone-based application. During the treatment phase, data from these recordings is used by an online therapist to make suggestions via text to the patient on the use of specific exercises within the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Current or previous former cancer diagnosis;
* Recurring cancer-related pain;
* Aged 18 years or older;
* Living in Sweden;
* Fluent in Swedish;
* Possession of a smartphone where they can download the application necessary for the daily diary recordings;
* Access to a device with internet access to receive the intervention;
* Not receiving another psychological treatment.

Exclusion Criteria:

- Not meeting any of the above inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain interference | From enrollment to the end of treatment at 6-8 weeks, and at month 5.
  The Brief Pain Inventory (BPI) scale was developed to assess the severity of pain and its impact on functioning. For the current study, the six questions assessing pain interference with daily activities will be used.
  Items will range from 0 to 100, with higher scores indicating worst outcomes. Only one of the items will be administered daily via a smart phone application.

SECONDARY OUTCOMES:
Pain severity | From enrollment to the end of treatment at 6-8 weeks, and at month 5.
  The Brief Pain Inventory (BPI) scale was developed to assess the severity of pain and its impact on functioning. For the current study, only 3 items will be used measuring pain severity at current, usual, and worst levels . Items will range from 0 to 100, with higher scores indicating worst outcomes. Only one of the items will be administered daily via a smart phone application.
Fatigue severity and interference | From enrollment to the end of treatment at 6-8 weeks, and at month 5.
  The Brief Fatigue Inventory (BFI) is a 9-item rating scale developed to assess subjective fatigue. The first three questions measure fatigue severity at current, usual, and worst levels. The following six questions assess fatigue interference with daily activities.
  Items will range from 0 to 100, with higher scores indicating worst outcomes. Only two of the items will be administered daily via a smart phone application.
Fear of cancer recurrence | From enrollment to the end of treatment at 6-8 weeks, and at month 5.
  The severity subscale of the Fear of Cancer Recurrence Inventory (FCRI) is used to assess fear of cancer recurrence. This 9-item subscale evaluates the presence and severity of intrusive thoughts associated with FCR. Each item is rated on a Likert scale ranging from 0 ("not at all" or "never") to 4 ("a great deal' or "all the time"), with higher scores indicating a worst outcome.
  Only two items will be administered daily via a smart phone application. These items will range from 0 to 100.
Depression | At enrollment, at month 2 and at month 5.
  The Patient Health Questionnaire (PHQ-9) is composed of 9 items that assess the frequency of depressive symptoms (feelings thoughts, states), from 0 ("Not at all) to 3 ("Nearly every day"), with higher scores indicating a worst outcome.
Anxiety | At enrollment, at month 2 and at month 5.
  The Generalised Anxiety Disorder-7 (GAD-7) scale is composed of 7 items that assess the different dimensions of the Generalised Anxiety Disorder and the patient is asked to mark the frequency of symptoms from 0 (='Never)' to 2 (='almost every day'), in the last two weeks. Higher scores indicate worst outcomes.
Well-being | At enrollment, at month 2 and at month 5.
  The Satisfaction with Life Scale (SWLS) is a 5-item scale designed to measure global life satisfaction, using a 7-point Likert scale, ranging from 1 (="strongly disagree") to 7 (=strongly agree), with higher scores indicating a better outcome.
Psychological flexibility | From enrollment to the end of treatment at 6-8 weeks, and at month 5.
  The Psy-Flex is a six-item self-report questionnaire assessing all six processes involved in ACT in a state form with high temporal specificity. Items are rated on a scale from 5 ("very often") to 1 ("very rarely"), with higher scores representing higher psychological flexibility.
  The Psychological Inflexibility (PI) subscale from the Multidimensional Psychological Flexibility Inventory (MPFI) measures the 5 dimensions of psychological inflexibility with responses given on a 6-point scale ranging from 1 (="never true) to 6 (="always true"), and with higher scores indicating higher levels of psychological inflexibility.
  Only the Psy-Flex will be administered daily via a smart phone application. These items will range from 0 to 100.
Overall functioning | Up to 6-8 weeks.
  One item measuring the physical ability to carry out daily activities ranging from 0 (=unable to carry out daily activities) to 100 (=able to carry out daily activities) will be used to assess overall functioning, with higher scores indicating better outcomes.
Mood | Up to 6-8 weeks.
  One item measuring mood, ranging from 0 (=negative) to 100 (=positive), with higher scores indicating better outcomes.
Subjective change | At month 2.
  The Patient Global Impression of Change (PGIC) scale is a single question asking respondents to rate how their condition has changed since the beginning of treatment, from 1 (=no change) to 7 (=a great deal better), with higher scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Perrin, PhD, Principal Investigator — Lund University
Locations (1):
- Lund University, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No